CLINICAL TRIAL: NCT04877873
Title: Dual-task Gait Performance in People With Knee Osteoarthritis Before and After Knee Replacement Surgery
Status: Completed | Type: Observational
Sponsor: University of Haifa (Other)
Collaborators: Emek Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: KneeOADualTask
Record Dates: First submitted 2021-05-02; First posted 2021-05-07 (Actual); Last update posted 2023-05-12 (Actual); Status verified 2022-05

CONDITIONS: Osteoarthritis, Knee
Keywords: Total knee replacement; Cognitive load; Gait; Proprioception; Dual task
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Postoperative Period

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No

INTERVENTIONS:
Behavioral: Gait analysis pre- and post- surgery — None (observational)

SUMMARY:
Knee Osteoarthritis (OA) is one of the most common conditions causing disability and limitation in the elderly population, with 13% of women and 10% of men over the age of 60 suffering from symptomatic knee osteoarthritis. Pain and other symptoms of OA significantly affect the quality of life, manifesting itself in pain, decreased range of motion, functional limitation and change in gait patterns.

Total Knee Replacement Surgery (TKR) is the most common solution for patients with advanced cartilage erosion and is considered a successful surgery with high satisfaction rates (about 80%). The surgery becomes necessary when pain limits the daily functioning and impairs the quality of life and after the failure of conservative treatment.

Still, patients undergoing TKR suffer in the first period after surgery from pain, decreased balance and proprioceptive impairment. Despite the improvement in pain and function, the rates of falls after surgery do not change drastically and remain high.

About a third of older adults fall each year, leading to fractures, functional decline and in some cases death. Walking is a complex task, and with advancing age walking becomes less automatic and requires additional attention. Among adults, it is known that an increased risk of falls is associated with reduced ability to perform complex walking tasks, such as walking while talking or crossing obstacles.

After TKR, most falls occur while walking due to slipping / tripping. In addition, proprioceptive impairment, pain and poor balance are associated with an increased risk of falling after TKR. The mechanism underlying these effects may be increased allocation of cognitive resources to walking. Thus, this study will examine the ability of people before and after TKR to perform complex walking tasks, in order to examine the change in attention allocation to walking following surgery. It is hypothesized that after surgery, the ability to walk while performing an additional task will be lower than prior to surgery.

ELIGIBILITY:
Inclusion Criteria:

* Able to walk at least for 1 minute with no assistive device
* Able to understand and complete simple instructions

Exclusion Criteria:

* Diagnosed dementia
* Diseases impairing balance
* Diagnosed rheumatoid arthritis

Ages: 65 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Candidates for TKR surgery at HaEmek Medical Center.
Sampling Method: Non-Probability Sample
Enrollment: 38 (Actual)
Dates: Start 2020-10-19 (Actual); Primary Completion 2022-08-01 (Actual); Study Completion 2022-08-01 (Actual)

PRIMARY OUTCOMES:
Change in Gait speed | One month prior to surgery, 4.5 months post-surgery
  Change in gait speed as measured using an instrumented mat
Change in gait variability | One month prior to surgery, 4.5 months post-surgery
  Change in coefficient of variation of stride time and stride length, as measured using an instrumented mat

SECONDARY OUTCOMES:
Change in Joint position sense | One month prior to surgery, 4.5 months post-surgery
  Estimation of knee position using the Physiological Profile Assessment (PPA). Specifically, the difference between intended knee flexion angle and achieved flexion angle is calculated in degrees (worse performance is identified via larger difference)
Change in Pain, stiffness, physical function | One month prior to surgery, 4.5 months post-surgery
  The Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Is a self-report questionnaire of pain, stiffness and physical function in people with knee osteoarthritis. Scores range 0-20 for pain, 0-8 for stiffness and 0-68 for physical function
Change in dynamic Balance | One month prior to surgery, 4.5 months post-surgery
  Mini Balance Evaluation Systems Test (Mini-BesTest) is a functional test of dynamic balance. Scores range from 0 to 28, with better scores indicating better balance.
Change in balance self-efficacy | One month prior to surgery, 4.5 months post-surgery
  The Activities-specific Balance Confidence (ABC) Scale is a self-reported measure of balance self-efficacy. Ranging from 0 to 100, better scores indicate better balance self-efficacy
Change in movement reinvestment | One month prior to surgery, 4.5 months post-surgery
  Movement reinvestment will be measured using the Movement Specific Reinvestment Scale (MSRS), a self-report measure of conscious monitoring of movement. Scores range from 10 to 60, with higher scores denoting more conscious movement monitoring
Cognitive function | One month prior to surgery
  Montreal Cognitive Assessment (MoCA) is a test of cognitive function. Ranging from 0 to 30, better scores denote better cognitive function.

CONTACTS AND LOCATIONS:
Locations (1):
- HaEmek Medical Center, Afula, Israel

IPD SHARING:
Plan to Share IPD: No